CLINICAL TRIAL: NCT06780163
Title: A Pre-Post Quasi-Experimental Study to Evaluate the Effects of Vaginal Estrogen on the Urine Microbiome and Overactive Bladder Symptoms in Menopausal Women
Brief Title: Effect of Vaginal Estrogen on Alterations in the Urine Microbiome of Menopausal Women With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MURA2024/948
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder (OAB); Menopause; Microbiome
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Estrogen (Experimental): Participants will receive 17β-estradiol vaginal tablets (10 mcg) daily for the first two weeks, followed by twice-weekly doses for a total of 12 weeks. Participants will be asked to bring the blister pack for pill count at the 12-week follow-up (checking for compliance)
  Interventions: Drug: 17β-estradiol 10 mcg

INTERVENTIONS:
Drug: 17β-estradiol 10 mcg — 17β-estradiol 10 mcg will be given to all participants. The participants will be asked to use 1 tab daily for 2 weeks vaginally before bed, then 1 tab twice a week vaginally before bed until 12 weeks
  Other Names: Femiest®

SUMMARY:
The goal of this Pre-Post Quasi-experimental study is to investigates the effect of vaginal estrogen therapy on changes in the urinary microbiome and its association with improvement in overactive bladder (OAB) symptoms in menopausal women

Primary Objective:

To evaluate the effects of vaginal estrogen on the level of Lactobacillus in the urine of postmenopausal women with OAB.

Secondary Objectives

1. To evaluate the effects of vaginal estrogen on urine microbiome in postmenopausal women with OAB.
2. To identify the association of alterations of urine microbiome after vaginal estrogen treatment with overactive bladder symptoms.

After informed and consents process, urine samples for microbiome study will be collected from participants with sterile technique. 17β-estradiol 10 mcg will be given to the participants. The participants will be ask to use 1 tab daily for 2 weeks vaginally before bed, then 1 tab twice a week vaginally before bed until 12 weeks. Then they will come back to hospital to take urine sample for microbiome study.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a common condition affecting 12-20% of adults, particularly women in the menopausal phase. OAB is characterized by urinary urgency, frequency, nocturia, and sometimes urgency urinary incontinence, significantly impairing quality of life. Menopause is associated with a decline in estrogen levels, which affects the integrity of the lower urinary tract and may contribute to OAB symptoms.

Vaginal estrogen therapy has been used to alleviate urogenital symptoms in postmenopausal women by improving vaginal atrophy, enhancing urethral closure pressure, and potentially improving bladder function. Recent studies have suggested that the urinary microbiome plays a critical role in urinary tract health and dysfunction. Alterations in the urinary microbiome, known as dysbiosis, have been linked to conditions such as OAB, urgency urinary incontinence, and recurrent urinary tract infections.

This pre-post quasi-experimental study aims to evaluate the effects of vaginal estrogen therapy on the urinary microbiome and its association with OAB symptom improvement in menopausal women. Specifically, the study will focus on:

1. Measuring changes in Lactobacillus abundance in urine after vaginal estrogen therapy. (Primary objective)
2. Measuring changes in the overall urinary microbiome diversity. (Secondary objective)
3. Identifying associations between changes in the microbiome and improvements in OAB symptoms. (Secondary objective)

The study will enroll 30 postmenopausal women with a clinical diagnosis of OAB who meet specific inclusion criteria. Participants will receive 17β-estradiol vaginal tablets (10 mcg) daily for the first two weeks, followed by twice-weekly doses for a total of 12 weeks. Urine samples will be collected via sterile catheterization at baseline and after 12 weeks to analyze microbiome diversity and Lactobacillus levels. OAB symptoms will be assessed using validated Thai versions of the Overactive Bladder Symptom Score (OABSS) and Overactive Bladder Questionnaire Short Form (OAB-q SF).

The findings from this study will provide valuable insights into the role of the urinary microbiome in the pathophysiology of OAB and the therapeutic effects of vaginal estrogen. This knowledge could pave the way for personalized treatments targeting hormonal and microbial factors in postmenopausal women with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Natural or surgical menopause at least 1 year
* Present with overactive bladder symptoms by using validated Thai version of OVERACTIVE BLADDER SYMPTOM SCORE (score in No.3 ≥ 2 and overall score ≥ 3)
* Absence of urinary infection
* Post-void residual urine less than 100ml

Exclusion Criteria:

* Currently or prior use of systemic hormone replacement therapy or vaginal estrogen within the past 3 months
* Contraindication or allergy to estrogen therapy
* Use of antibiotics, prebiotics and probiotics within the past 2 weeks
* Currently on antimuscarinic or β3 agonists medication or within the past 3 months
* Pelvic organ prolapse greater than stage II

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Lactobacillus abundance | From enrollment to the end of treatment at 12 weeks
  Change in Lactobacillus abundance (measure by urine microbiome study) after vaginal estrogen therapy

SECONDARY OUTCOMES:
Change in urine microbiome diversity | From enrollment to the end of treatment at 12 weeks
  Change in urine microbiome diversity after vaginal estrogen therapy (measured by urine microbiome study)
Association of change in urine microbiome with overactive bladder symptoms | From enrollment to the end of treatment at 12 weeks
  Association of change in urine microbiome with overactive bladder symptoms measured by questionnaire (OAB-q SF)

CONTACTS AND LOCATIONS:
Overall Officials: Jittima Manonai, MD, Study Chair — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared in de-identified data.
  Research collaborators will have access to the data.
  Specify that data shared with collaborators will be used for conducting analyses relevant to the study objectives, secondary analyses, or other agreed-upon purposes.
  Data will be shared via a secure institutional repository accessible to collaborators through data-sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared with research collaborators upon completion of the primary analysis and will remain accessible for 5 years after the study's conclusion.
Access Criteria: Only research collaborators will have access to the data.

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Weber MA, Kleijn MH, Langendam M, Limpens J, Heineman MJ, Roovers JP. Local Oestrogen for Pelvic Floor Disorders: A Systematic Review. PLoS One. 2015 Sep 18;10(9):e0136265. doi: 10.1371/journal.pone.0136265. eCollection 2015. PMID 26383760
- [Background] Krause M, Wheeler TL 2nd, Snyder TE, Richter HE. Local Effects of Vaginally Administered Estrogen Therapy: A Review. J Pelvic Med Surg. 2009 May;15(3):105-114. doi: 10.1097/SPV.0b013e3181ab4804. PMID 22229022
- [Background] Cardozo LD, Wise BG, Benness CJ. Vaginal oestradiol for the treatment of lower urinary tract symptoms in postmenopausal women--a double-blind placebo-controlled study. J Obstet Gynaecol. 2001 Jul;21(4):383-5. doi: 10.1080/01443610120059941. PMID 12521832
- [Background] Simunic V, Banovic I, Ciglar S, Jeren L, Pavicic Baldani D, Sprem M. Local estrogen treatment in patients with urogenital symptoms. Int J Gynaecol Obstet. 2003 Aug;82(2):187-97. doi: 10.1016/s0020-7292(03)00200-5. PMID 12873780
- [Background] Gasiorek M, Hsieh MH, Forster CS. Utility of DNA Next-Generation Sequencing and Expanded Quantitative Urine Culture in Diagnosis and Management of Chronic or Persistent Lower Urinary Tract Symptoms. J Clin Microbiol. 2019 Dec 23;58(1):e00204-19. doi: 10.1128/JCM.00204-19. Print 2019 Dec 23. PMID 31619534
- [Background] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT06780163/Prot_SAP_000.pdf